CLINICAL TRIAL: NCT06382272
Title: Bionic Breast Project: A Neuroprosthesis to Restore Touch Sensation and Reduce Chronic Pain After Mastectomy
Brief Title: A Bionic Breast Project Using Neuroprosthesis to Reduce Chronic Pain After Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB23-2027
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Mastectomy; Breast; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Mastectomy/Reconstruction (Experimental): Standard treatment our intervention/arm is just the implanting of the device.
  Interventions: Device: Bionic Breast implant

INTERVENTIONS:
Device: Bionic Breast implant — A small medical device will be temporarily implanted in one of the breasts at the time of the mastectomy. This device is capable of sending very small electrical currents to the nerves that can deliver sensory stimulation in response to touch and pressure applied to the breast

SUMMARY:
This trial seeks to establish whether or not touch sensation can be restored to the breast via neural stimulation. Data will also be obtained to inform future feasibility (including safety), efficacy, and acceptability trials.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Scheduled for bilateral mastectomy with two-stage (tissue expander) reconstruction at UCM
* Bilateral mastectomy for unilateral in situ or T1 (<2 cm), N0 (no lymph node involvement) breast cancer or breast cancer risk reduction due to known elevated breast cancer risk. (Note - 19-34% of women choosing mastectomy for small unilateral breast cancer elect bilateral mastectomy.)40 We will enroll from this cohort.
* Agrees to have breast tissue expander removed within 12-20 weeks of implantation.
* Has access to a cell phone and willing to provide the research interviewer with the cell phone number
* Agrees to receive text messages from the study
* Able to speak and understand English or Spanish
* Able to participate in the informed consent process

Exclusion criteria:

* Requires breast radiation
* Single stage mastectomy and reconstruction procedure
* Clinical evidence of bilateral breast cancer
* Clinical evidence of lymph node involvement
* Prior history of mastectomy or other major breast surgery
* Prior history of radiation to the chest area (e.g., mantle radiation for Hodgkin's disease)
* Prior history of injury (e.g., trauma, surgery, burn) that the participant perceives to have had an effect on the sensation of the breast
* Pregnant or intending to become pregnant during the study period
* Pacemaker, defibrillator or other implanted electrical stimulation device that may be affected by the implanted electrodes
* Complex regional pain syndrome or other pain syndromes or a history of a neurologic condition like multiple sclerosis, degenerative neurological disease, cognitive impairment or dementia
* Uncontrolled diabetes
* History of poor wound healing or chronic skin ulcerations
* History of uncontrolled infection or active infection at time of consent
* Expectation that MRI will be required while the devices are implanted
* Inability or unwillingness to follow verbal instructions and comply with study procedures
* Untreated or poorly managed physical or mental health condition that may pose additional risk according to clinical judgment of the patient's breast surgeon or surgeons
* Unwillingness to undergo psychological evaluation to determine study eligibility, if requested or required by surgeons or investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychophysical tasks to assess stimulation-elicited sensation | 7 months after mastectomy+implantation and removal of device
  The purpose of the detection task is to determine the minimum pulse amplitude (PA) required to elicit a detectable percept for each C-FINE contact.

SECONDARY OUTCOMES:
Maximum stimulation level | 7 months after mastectomy+implantation and removal of device
  To determine the maximum range of stimulation that elicits comfortable sensation.
Amplitude discrimination task | 7 months after mastectomy+implantation and removal of device
  The purpose of this task is to determine the amount by which PA needs to be changed to evoke a reliably distinguishable percept for each C-FINE contact.
Frequency discrimination task | 7 months after mastectomy+implantation and removal of device
  The purpose of this task is to determine the amount by which pulse frequency (PF) needs to change to evoke a reliably distinguishable percept for each C-FINE contact.
Magnitude estimation | 7 months after mastectomy+implantation and removal of device
  The purpose of this task is to (further) characterize the relationship between PA/PF and sensory magnitude.
Projected field mapping | 7 months after mastectomy+implantation and removal of device
  The purpose of this task is to map the location of percepts evoked by stimulation through each C-FINE contact.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Lindau, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No